CLINICAL TRIAL: NCT01740271
Title: Pharmacogenetic Dosing of Epirubicin in FEC Chemotherapy
Brief Title: A Study of Genetic Based Chemotherapy Dosing for Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEC100-01
Record Dates: First submitted 2012-11-16; First posted 2012-12-04 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; non-metastatic carcinoma of the breast chemotherapy; adjuvant therapy; neoadjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epirubicin (Experimental): Following genetic analysis, depending on results, participants will receive either standard or increased epirubicin dosing for cycles 2 - 4.
  Interventions: Drug: Epirubicin

INTERVENTIONS:
Drug: Epirubicin

SUMMARY:
Epirubicin is a common chemotherapy medication used in the treatment of breast cancer. However, chemotherapy dosing is calculated based on people's height and weight, which may not be the most accurate way. The purpose of this study is to see if epirubicin dosing based on people's genetic profiles is better than the usual methods.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with histologically confirmed non-metastatic invasive breast cancer who are scheduled to receive at least three cycles of FEC100 in the adjuvant or neoadjuvant setting
2. Documented pathological evaluation of the breast cancer for hormone receptor (estrogen receptor [ER], progesterone receptor [PR] and HER-2 status
3. Eastern Cooperative Oncology (ECOG) performance status of ≤ 2
4. A Left Ventricular Ejection Fraction (LVEF) ≥ 50%.

Exclusion Criteria:

1. Uncontrolled congestive heart failure (CHF) or angina, history of myocardial infarction within 2 months before study enrollment, or cardiac functional capacity Class III or IV as defined by the New York Heart Association Classification.
2. Psychiatric disorder(s) that would interfere with consent, study participation, or follow up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The goal of this study is to determine the safety of pharmacogenetic guided dosing of epirubicin for each UGT2B7 genotype. | 10 years
  Primary Objectives To describe the side effects of pharmacogenetically individualized FEC chemotherapy in the adjuvant and neoadjuvant treatment of breast cancer.

SECONDARY OUTCOMES:
Secondary Objectives i) To verify relationships between uridine glucuronosyltransferase 2B7 polymorphisms and epirubicin pharmacokinetics ii) To verify relationships between body composition and epirubicin pharmacokinetics | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Sawyer, MD FRCPC BScPharm, Principal Investigator — Alberta Health services; John R Mackey, MD FRCPC, Study Director — Alberta Health services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada